CLINICAL TRIAL: NCT03159663
Title: Assessment of Quality of Life in Hemophiliac Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, peter khalil, assiut, Assiut University
Other Study IDs: Assiut1987
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Improvement of Quality of Life of Hemophiliac Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Hemophilia is an X-linked congenital bleeding disorder caused by deficiency of coagulation factor VIII (in hemophilia A) or factor IX (in hemophilia B).

The deficiency is the result of mutations of the respective clotting factor genes.

DETAILED DESCRIPTION:
Hemophilia is rare, with only about 1 instance in every 10,000 births (or 1 in 5,000 male births) for hemophilia A and 1 in 50,000 births for hemophilia B.

According to the World Federation of Hemophilia, 400 000 people worldwide & 5,307 people in Egypt are suffering from hemophilia.

Hemophilia A is more common than hemophilia B, representing 80-85 % of the total hemophilia population.

Signs and symptoms of hemophilia vary according to the level of clotting factors, mild, moderate and sever.

* Unexplained excessive bleeding from cuts or injuries
* Epistaxis without a known cause
* Many large or deep bruises
* Hamoarthritis
* Hematuria and Melena.
* Intracranial hemorrhage and death
* In infants, unexplained irritability

it is subjective representation of health, including not only physical,mental and social, but also emotional and everyday life dimensions in terms of well-being. Several definitions of QoL have been provided, the definition of the WHO viewing QoL as 'individuals perceptions of their position in life in the context of culture and value systems in which they live and in relation to their goals, expectation standards and concerns'

ELIGIBILITY:
Inclusion Criteria:

* - Hemophilia A & B
* Different age groups (pediatric - adolescence - adult )
* Home or hospitalized treatment
* complications such as joint swelling , spontaneous bleeding, etc….

Exclusion Criteria:

- 1- Other causes of bleeding tendency such as liver failure, DIC, anticoagulant drugs, etc..

2- Diseases that affect joints such as osteoarthritis, SLE , etc.. 3- Mentally retarded patients.

Ages: 10 Years to 70 Years | Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: all patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2017-06-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
evaluation and improvement of quality of life of hemophiliac patients | one year
  by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided